CLINICAL TRIAL: NCT04690426
Title: A Phase 1, First-in-Human, Randomized, Double-Blind, Placebo-Controlled, Multiple-Dose-Escalation Study to Evaluate the Safety, Tolerability, and Immunogenicity of PRV-101, a Coxsackie Virus B (CVB) Vaccine, in Healthy Adult Subjects
Brief Title: PROtocol for Coxsackievirus VaccinE in Healthy VoluNTteers
Acronym: PROVENT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Provention Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: PRV-101-001
Record Dates: First submitted 2020-12-15; First posted 2020-12-30 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Viral; Infection, Coxsackie(Virus)
Keywords: Coxsackie Virus B, vaccine
MeSH Terms: conditions — Coxsackievirus Infections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Cohort 1, Low Dose, Placebo (Placebo Comparator): Low dose of placebo by intramuscular injection, 3 doses at 4-week intervals
  Interventions: Other: Placebo
- Cohort 1, Low Dose, PRV-101 (Experimental): Low dose of PRV-101 by intramuscular injection, 3 doses at 4-week intervals
  Interventions: Biological: PRV-101
- Cohort 2, High Dose, Placebo (Placebo Comparator): High dose of placebo by intramuscular injection, 3 doses at 4-week intervals
  Interventions: Other: Placebo
- Cohort 2, High Dose, PRV-101 (Experimental): High dose of PRV-101 by intramuscular injection, 3 doses at 4-week intervals
  Interventions: Biological: PRV-101

INTERVENTIONS:
Biological: PRV-101 — Coxsackie Virus B vaccine
  Arms: Cohort 1, Low Dose, PRV-101; Cohort 2, High Dose, PRV-101
Other: Placebo — Placebo
  Arms: Cohort 1, Low Dose, Placebo; Cohort 2, High Dose, Placebo

SUMMARY:
Phase 1, first-in-human, randomized, double-blind, placebo-controlled, multiple-dose-escalation study to evaluate the safety, tolerability and immunogenicity of PRV-101, a coxsackie virus B vaccine, in healthy volunteers.

DETAILED DESCRIPTION:
Thirty two healthy adult subjects will be enrolled into 2 dose cohorts (low-dose and high-dose cohorts, 16 subjects per cohort) and will be randomized in a double-blind manner to PRV-101 or placebo in a 3:1 ratio. Each subject will receive up to 3 administrations of the study drug (PRV-101 or placebo) at 4-week intervals and will be followed for 24 weeks after the final dose. Each cohort will start with a sentinel dosing group (2 subjects). Cohort 2 will commence after safety data from the first 2 doses from all Cohort 1 participants are reviewed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults, males and females, ages 18 to 45 yrs, with BMI 19 to 30 kg/m2
* Women of childbearing potential must have negative pregnancy test and agree to use an acceptable method of highly effective contraceptive
* Men must either have a vasectomy or agree to use highly effective contraception

Exclusion Criteria:

* Prior or current clinically significant medical illness or disorder
* Has celiac disease or type 1 diabetes or related autoantibodies
* Has active acute or chronic/latent infection, or history of recent serious infection
* Recent acute illness or recent major illness, hospitalization or surgery
* Recent history of alcohol or drug abuse
* Received an experimental antibody or biologic therapy in last 6 months
* Received live, inactivated or subunit virus vaccine or a bacterial vaccine within last 4 weeks
* Intolerance or hypersensitivity to vaccines or vaccine components or has a drug or food allergy or allergic disease requiring medication

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-12-07 (Actual); Study Completion 2021-12-07 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events (safety and tolerability) | Throughout the 32 weeks of the study
  Adverse events will be assessed by frequency and criteria for severity (mild, moderate or severe)

SECONDARY OUTCOMES:
Development of neutralizing antibodies to coxsackie B virus (immunogenicity, efficacy) | Days 1, 29, and 57 and Weeks 12 and 32
  Proportion of responders (ie, those that seroconvert or have at least a 4-fold increase in neutralizing antibody titers to any of the coxsackie B virus strains as measured by plaque reduction assay using serial serum dilutions)
Titer of antibodies to coxsackie B virus (immunogenicity, efficacy) | Days 1, 29 and 57 and weeks 12 and 32
  Mean and peak geometric mean serum IgG titers of antibodies against any of the coxsackie B virus strains, measured by ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Chief Scientific Officer, Principal Investigator — CRST Oy
Locations (1):
- Clinical Research Services Turku (CRST) Oy, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hyoty H, Kaariainen S, Laiho JE, Comer GM, Tian W, Harkonen T, Lehtonen JP, Oikarinen S, Puustinen L, Snyder M, Leon F, Scheinin M, Knip M, Sanjuan M. Safety, tolerability and immunogenicity of PRV-101, a multivalent vaccine targeting coxsackie B viruses (CVBs) associated with type 1 diabetes: a double-blind randomised placebo-controlled Phase I trial. Diabetologia. 2024 May;67(5):811-821. doi: 10.1007/s00125-024-06092-w. Epub 2024 Feb 19. PMID 38369573